CLINICAL TRIAL: NCT03704077
Title: A Randomized, Active-Controlled, Open-Label, Phase 2 Clinical Trial of BMS-986213, in Combination With Various Standard-of-Care Therapeutic Regimens, in Participants With Recurrent, Locally Advanced, or Metastatic Gastric Cancer (GC) or Gastroesophageal Junction (GEJ) Adenocarcinoma
Brief Title: An Investigational Immuno-therapy Study of Relatlimab Plus Nivolumab Compared to Various Standard-of-Care Therapies in Previously Treated Participants With Recurrent, Advanced or Metastatic Gastric Cancer or Gastroesophageal Junction Adenocarcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Replaced it with another clinical trial
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA224-061; 2018-001070-20 (EudraCT Number)
Record Dates: First submitted 2018-10-09; First posted 2018-10-12 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Gastric Cancer; Cancer of the Stomach; Stomach Cancer; Gastroesophageal Junction
MeSH Terms: conditions — Stomach Neoplasms | interventions — relatlimab; Nivolumab; Paclitaxel; Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort A: relatlimab + nivolumab + paclitaxel (Experimental)
  Interventions: Biological: Relatlimab + Nivolumab; Biological: Nivolumab; Drug: Paclitaxel
- Cohort A: nivolumab + paclitaxel (Experimental)
  Interventions: Biological: Nivolumab; Drug: Paclitaxel
- Cohort A: ramucirumab + paclitaxel (Active Comparator): Standard-of-care
  Interventions: Drug: Paclitaxel; Drug: Ramucirumab
- Cohort B: relatlimab + nivolumab (Experimental)
  Interventions: Biological: Relatlimab + Nivolumab; Biological: Nivolumab
- Cohort B: nivolumab (Active Comparator): Standard-of-care
  Interventions: Biological: Nivolumab
- Cohort C: relatlimab + nivolumab (Experimental)
  Interventions: Biological: Relatlimab + Nivolumab; Biological: Nivolumab

INTERVENTIONS:
Biological: Relatlimab + Nivolumab — Specified dose on specified days
  Other Names: BMS-986213
  Arms: Cohort A: relatlimab + nivolumab + paclitaxel; Cohort B: relatlimab + nivolumab; Cohort C: relatlimab + nivolumab
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo
  Arms: Cohort A: nivolumab + paclitaxel; Cohort A: relatlimab + nivolumab + paclitaxel; Cohort B: nivolumab; Cohort B: relatlimab + nivolumab; Cohort C: relatlimab + nivolumab
Drug: Paclitaxel — Specified dose on specified days
  Other Names: Taxol; Onxal
  Arms: Cohort A: nivolumab + paclitaxel; Cohort A: ramucirumab + paclitaxel; Cohort A: relatlimab + nivolumab + paclitaxel
Drug: Ramucirumab — Specified dose on specified days
  Other Names: Cyramza
  Arms: Cohort A: ramucirumab + paclitaxel

SUMMARY:
The purpose of this study is to determine the effectiveness of relatlimab plus nivolumab, alone or in combination with various standard-of-care treatments in participants with gastric cancer (GC) or gastroesophageal junction (GEJ) adenocarcinoma that has come back or spread to other places in the body after prior therapy.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced or recurrent or metastatic GC or GEJ adenocarcinoma that is considered incurable by local therapies such as radiation or surgery
* Evidence of progressive disease (PD) on at least one prior platinum- and fluoropyrimidine-containing chemotherapy regimen
* Available tumor tissue for biomarker analysis

Exclusion Criteria:

* Must not have squamous cell or undifferentiated GC or GEJ
* Untreated known central nervous system (CNS) metastases
* Uncontrolled or significant cardiovascular disease

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-31 (Estimated); Primary Completion 2022-02-27 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Approximately 31 months

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Approximately 5 years
Incidence of serious adverse events (SAEs) | Approximately 5 years
Incidence of AEs leading to discontinuation | Approximately 5 years
Incidence of deaths | Approximately 5 years
Incidence of laboratory abnormalities | Approximately 5 years
ORR | Approximately 5 years
  Cohort A1
Duration of response (DOR) | Approximately 5 years
Progression free survival (PFS) | Approximately 5 years
Overall survival (OS) | Approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (79):
- United States (20):
  - Local Institution, Daphne, Alabama
  - Local Institution, Bakersfield, California
  - Local Institution, Fullerton, California
  - Local Institution, Los Angeles, California
  - Local Institution, Redondo Beach, California
  - Local Institution, Santa Barbara, California
  - Local Institution, Aurora, Colorado
  - Local Institution, Lakewood, Colorado
  - Local Institution, Miami, Florida
  - Local Institution, Tampa, Florida
  - Local Institution, Marietta, Georgia
  - Local Institution, Boston, Massachusetts
  - Local Institution, St Louis, Missouri
  - Local Institution, New Brunswick, New Jersey
  - Local Institution, Chapel Hill, North Carolina
  - Local Institution, Charlotte, North Carolina
  - Local Institution, Fargo, North Dakota
  - Local Institution, Allentown, Pennsylvania
  - Local Institution, Sioux Falls, South Dakota
  - Local Institution, Vancouver, Washington
- Argentina (4):
  - Local Institution, Viedma, Río Negro Province
  - Local Institution, Buenos Aires
  - Local Institution, CABA
  - Local Institution, Córdoba
- Australia (6):
  - Local Institution, Westmead, New South Wales
  - Local Institution, Heidelberg, Victoria
  - Local Institution, Malvern, Victoria
  - Local Institution, Melbourne, Victoria
  - Local Institution, Bedford Park
  - Local Institution, Murdoch
- Brazil (7):
  - Local Institution, Fortaleza, Ceará
  - Local Institution, Belo Horizonte, Minas Gerais
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Barretos, São Paulo
  - Local Institution, Jaú, São Paulo
  - Local Institution, Rio de Janeiro
  - Local Institution, São Paulo
- Canada (6):
  - Local Institution, Halifax, Nova Scotia
  - Local Institution, Hamilton, Ontario
  - Local Institution, Ottawa, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Montreal, Quebec
  - Local Institution, Sherbrooke, Quebec
- Local Institution, Santiago, Santiago Metropolitan, Chile
- Local Institution, Medellín, Colombia
- Germany (15):
  - Local Institution, Berlin
  - Local Institution, Cologne
  - Local Institution, Erlangen
  - Local Institution, Essen
  - Local Institution, Frankfurt am Main
  - Local Institution, Freiburg im Breisgau
  - Local Institution, Hamburg
  - Local Institution, Hanover
  - Local Institution, Jena
  - Local Institution, Mainz
  - Local Institution, Mannheim
  - Local Institution, Marburg
  - Local Institution, Paderborn
  - Local Institution, Reutlingen
  - Local Institution, Wiesbaden
- Italy (4):
  - Local Institution, Bergamo
  - Local Institution, Milan
  - Local Institution, Napoli
  - Local Institution, Reggio Emilia
- Mexico (5):
  - Local Institution, Tuxtla Gutiérrez, Chiapas
  - Local Institution, ZONA Centro. LEON, Guanajuato
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Mérida, Yucatán
  - Local Institution, Aguascalientes
- Portugal (2):
  - Local Institution, Lisbon
  - Local Institution, Porto
- Local Institution, Rio Piedras, Puerto Rico
- Romania (4):
  - Local Institution, Bucharest
  - Local Institution, Cluj-Napoca
  - Local Institution, Craiova
  - Local Institution, Floreşti
- Spain (3):
  - Local Institution, Badajoz
  - Local Institution, Madrid
  - Local Institution, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Individual patient level data from this study may be shared with qualified researchers, upon request, following the timelines and process detailed on https://www.bms.com/researchers-and-partners/independent-research/data-sharing-request-process.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm